CLINICAL TRIAL: NCT02068066
Title: Physical Workload and Work Capacity Across Occupational Groups
Status: Completed | Type: Observational
Sponsor: Cantonal Hosptal, Baselland (Other)
Collaborators: Swiss National Accident Insurance Institution (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Jörg Leuppi, Head of Medical University Clinic, Cantonal Hosptal Baselland, Cantonal Hosptal, Baselland
Other Study IDs: 260/12
Record Dates: First submitted 2014-02-19; First posted 2014-02-20 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Occupational Rehabilitation; Professional Reintegration; Work Load; Work Capacity
Keywords: Physical work requirements; Energy expenditure; Physical activity; Different occupational categories; Aerobic capacity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Physical activity is defined as any bodily movement produced by skeletal muscles resulting in energy expenditure (Caspersen, 1985). According to classical work physiology, energy expenditure was considered as basis for assessing the severity of manual work (Grandjean 1991). Steele et. al. found blue collar workers to report significantly more walking activity, daily step counts and MET min/week than professionals and white collar workers. However, the energy cost of physical activity may not necessarily be equivalent to body movement. Therefore, modern concepts include also other aspects reflecting the amount of workload. Soer et. al. applied an evaluation system consisting 12 work-related tests to establish functional capacity in healthy employees. The assessment included various lifting and energetic tasks as well as coordination exercises. In occupational rehabilitation a balance between workload and work capacity is necessary for professional reintegration. Thus, it is of great value to evaluate a wide range of work requirements across occupational groups in terms of energy expenditure, physical activity and aerobic capacity.

Aim: The aim of this study is to examine the amount of physical activity and energy expenditure during a normal working day with focus on differences between occupational groups.

Method: To analyze the situation in Switzerland, 300 healthy and full-time employed adults between 18-65 years will be investigated in the Basel region. Participants will be stratified by occupational category according to the ISCO-88 and will then be merged into 3 groups with low-, moderate- and high-intensity occupational activity. By wearing the SenseWear Mini Armband on 7 consecutive days, average daily energy expenditure, activity duration at different intensities and step counts will be assessed during work-time. In addition, individual's aerobic capacity will be determined by the 20-meter shuttle run test.

Outlook: This study is expected to provide detailed information about physical work requirements with regard to professional reintegration. For developing adequate intervention and treatment strategies, it is of great value to evaluate performance criteria across occupational groups.

DETAILED DESCRIPTION:
1. Introduction

   1.1 Background

   Regarding occupational rehabilitation, a balance between workload and individual's work capacity is required for returning to work successfully after an injury or illness. Therefore, it is of great value to evaluate a wide range of physical work requirements and to assess employee's work capacity across occupational groups. Although several approaches have been made in this regard, there are few objective data available so far and no established reference values exist to evaluate, whether, when and how a return to work is possible. One reason could be that objectifying workload and work capacity is methodically challenging because of their multidimensional nature [1, 2].

   Physical activity is defined as any bodily movement produced by skeletal muscles resulting in energy expenditure [3]. In classical work physiology, energy expenditure was therefore considered as basis for assessing the amount of workload [4, 5]. However, the energy cost of physical activity may not necessarily be equivalent to body movement [6]. For that reason, modern concepts include also other aspects reflecting the severity of manual work. The 'Dictionary of Occupational Titles' (DOT), developed by the U.S. government, classifies professions into five categories (sedentary, light, medium, heavy, very heavy) based on the amount of energy expended as well as on the intensity and duration of lifting or carrying during work [7]. Though, the DOT classification has not been based on quantitative work-related analyses, but rather on consensus meetings of experts. Furthermore, its validity has not been established.

   Work capacity can be assessed using functional capacity evaluations (FCEs), which measure the ability of subjects to perform specific activities [8]. Worldwide, there are various FCE protocols available being job specific [9], pathology specific [10, 11] or of a more general type. Soer et al. applied an evaluation system consisting of 12 work-related tests to establish functional capacity in healthy employees [12]. The assessment included various lifting and energetic exercises as well as coordination tasks. From the test results, normative FCE values were acquired for each DOT-category, which can be compared to patient data in order to make work recommendations.

   However, since validity of the DOT has not been proved, further analysis concerning workload assessment is required. Moreover, the application of such complex FCE tools is related to high expenses and efforts and may therefore not be appropriate in a general clinical or field context. Especially in large populations, implementing highly accurate instruments is difficult due to high costs and poor practicability [13].

   For these reasons, the present study will focus on workload by investigating a wide range of physical work requirements across occupational groups and putting them in relation to employees' aerobic capacity. Since physical activity is characterized by various dimensions, such as duration and intensity [3], these factors will be considered for a comprehensive analysis.

   1.2 Specific aims

   The primary aim of this study is to investigate healthy employees in Switzerland regarding energy expenditure, metabolic equivalents (METs), physical activity duration at different intensities and the number of steps taken during a normal working day with focus on differences between occupational groups. Furthermore, the association between physical activity and aerobic capacity will be examined.

   1.3 Hypotheses

   1.3.1 Individuals practising heavy work are more physically active and consume more energy than those with light work.

   1.3.2 Aerobic capacity (VO2max) correlates positively with work and non-work related physical activity.

   1.4 Potential significance

   This study is expected to provide detailed information about physical work requirements and performance criteria of different occupational groups. This may be valuable regarding treatment and professional reintegration after an injury or illness, since up to now no established reference values exist. Objective workload data might improve intervention strategies and clinicians' recommendations for a successful return to work.
2. Methods

   2.1 Study design

   2.1.1 Primary and secondary outcomes

   Our primary objective is to analyze work related physical activity parameters measured by the SenseWear Mini armband and aerobic capacity determined by the 20-meter shuttle run test across occupational groups. Furthermore, perceived work intensity, activity behaviour in recreation, quality of life, body composition and several personal- and job-related factors will be investigated as secondary outcomes.

   2.1.2 Study procedures

   In this cross-sectional study, we plan to recruit healthy and full-time employed adults from different occupational fields in the Basel region, Switzerland. It is intended to start with a pilot study in January 2013, in which a total of 15 persons will be examined.

   Recruitment will initiate in May 2013 and will end as soon as 300 individuals are included in the study.

   Potential subjects will be contacted and asked for study participation by phone or by mail. Willing individuals meeting the inclusion criteria will fill out the informed consent form before starting the measurement procedure.

   At the first study visit, body measurements will be carried out such as height, weight and waist circumference (WC) and body mass index (BMI) will be calculated. In addition, a variety of personal- and job-related factors will be recorded. Furthermore, subjects will perform a 20-meter shuttle run in order to measure aerobic capacity.

   During the subsequent week, participants will be instructed to document their daily work activities and to rate their work related physical exertion twice per day using the Borg Scale. Moreover, by wearing the SenseWear Mini armband on seven consecutive days, physical activity and energy expenditure will be objectified.

   One week later at the second study visit, all subjects will complete several self-administered questionnaires concerning work and non-work related physical activity behaviour (IPAQ), health-related quality of life (SF-36) and self-assessment of professional activity and its intensity (VAS). In addition, open questions will be asked to each participant about past-week physical exertion in comparison to a normal week.

   The time required for the two study visits taking place at the individual's workstation, will be around 90 minutes per person. In addition, every participant will wear the activity monitor on seven consecutive days.

   Termination criteria for the measurements are skin irritations caused by the SenseWear Mini armband and exertional dyspnea during 20-meter shuttle run.

   2.2 Selection of study participants

   2.2.1 Recruitment

   In this study, it is intended to recruit 300 subjects from different occupational groups with low-, moderate- and high-intensity occupational activity, which are defined in a later section (see chapter 2.3.2). Based on this classification, companies will be selected. In each occupational group, 100 participants will be enrolled. Furthermore, homogeneity of age and gender within each group will be aimed at recruiting.

   First, we will contact the management of potential enterprises in order to present our project. If they are interested in a collaboration, we will ask for contact details of potentially recruitable employees, who will then be addressed by a member of our research team. Individuals will be informed and asked for study participation by phone or by email. Furthermore, it is planned to distribute study flyers in the companies, so that interested employees have the opportunity to contact us directly. In both situations, the recruitment and information process will be done externally.

   2.2.2 Inclusion criteria

   Healthy and full-time employed individuals between the age of 18 and 65, who have a sufficient knowledge of the German language in order to fill in the self-administered questionnaires by themselves.

   2.2.3 Exclusion criteria

   Subjects not giving consent for participation as well as those with movement restrictions, various diseases and accidents within the last three months that affect productivity at the workplace, cannot take part in this study. Furthermore, night shift workers will be excluded from participation.

   2.3 Instruments

   2.3.1 Personal- and job-related factors

   For each subject, gender (male / female) and employment (temporary / permanent) will be assessed as binary variables. Nationality (Swiss / EU / other), marital status (single / married / divorced) and smoking status (yes / no / never) will be recorded with three categories, while alcohol consumption (never / once to several times per month / once to several times per week / once per day), German skills (very good / good / medium / bad / very bad), highest education (compulsory school / apprenticeship / higher vocational school / diploma or maturity / university) and working time model (flextime / fix time / shift work / weekend work) will be evaluated with four, five and six categories, respectively. Age, native language, profession, avocation, medication, illnesses, accidents and working hours will be asked as open questions. Furthermore, to get an overview of the individual work activity, participants will be asked to keep a daily list of the main completed tasks including time information in accordance with the questionnaire regarding professional integration and pension [14].

   2.3.2 Classification of occupations

   The reported professions will be classified into 9 categories based on the International Standard Classification of Occupations ISCO-88 [15] (1. Managers, 2. Scientists, 3. Technicians, 4. Office workers, 5. Service workers, 6. Agricultural workers, 7. Craftsmen, 8. Machine operators, 9. Labourers). These 9 categories will then be collapsed into 3 groups with low-, moderate-and high-intensity occupational activity according to Suva experts in the field of ergonomics (1st group: Categories 1 (Managers), 2 (Scientists) and 4 (Office workers); 2nd group: Categories 3 (Technicians), 5 (Service workers) and 8 (Machine operators); 3rd group: Categories 6 (Agricultural workers), 7 (Craftsmen) and 9 (Labourers). Reliability of this stratification has been previously shown [16, 17].

   2.3.3 International Physical Activity Questionnaire

   The International Physical Activity Questionnaire (IPAQ) represents a convenient and simple instrument for measuring health enhancing physical activity at the population level. The self-administered long version of the IPAQ, being freely available in internet [18], will be used in the present study. It includes 26 questions and assesses past-week frequency (days) and duration (time per day) of physical activity within the domains of work, leisure-time, transport, domestic and garden. Moreover, each domain consists of walking, moderate and vigorous activities.

   According to the IPAQ guidelines for data analysis [19], continuous scores in form of MET-minutes per week will be calculated for each domain. MET-minutes per week, defined as energy costs of physical activity, will be computed by multiplying the intensity (specific MET value) of an activity with its frequency (days) and duration (minutes). The corresponding MET values are set by the IPAQ guidelines based on the compendium of physical activity [20].

   According to numerous validity and reliability tests carried out in twelve different countries, the IPAQ is considered as an internationally valid assessment tool with acceptable measurement properties [21]. The long version of the IPAQ was translated into German as part of a dissertation and was validated in an Austrian sample [22]. It could be shown that it is suitable for research purposes with regard to physical activity detection [23].

   2.3.4 SF-36

   The SF-36 is a general quality of life questionnaire consisting of 36 items, which are formatted as binary questions or as semantic six-point differential scales. It refers to the past four weeks and includes nine content areas concerning vitality, general health perception, physical functioning, social functioning, role limitations (emotional/physical problems), pain, mental health and health change [24]. The SF-36 is considered to be the gold standard for measuring functional status and health-related quality of life and is therefore the most used questionnaire in this context [25].

   Since physical and mental disorders as well as pain may influence activity behaviour, the SF-36 will be used in the present study to adjust for potential confounders.

   2.3.5 Visual Analogue Scale

   The Visual Analogue Scale (VAS) is a measuring instrument for subjective characteristics that cannot be directly measured. Individuals express their response to a VAS item by marking a position along a continuous line between two end-points.

   The indicated locus will then be quantified by a defined scale [26]. In epidemiologic and clinical research, the most common VAS is a straight horizontal line of 100 mm length with its ends representing extreme limits of the measured parameter (worst - best) [27]. The VAS score is determined by measuring the distance in mm from the left end of the line to the point marked by the participant. Validity and reliability of VAS have been scientifically tested for a variety of parameters, such as acute and chronic pain [28, 29].

   In this study, individual's perception of past-week work and non-work related physical exertion and effort will be assessed by 100mm VASs. This may be valuable to evaluate whether the investigated period (exposure time) is representative and reflects a normal week.

   2.3.6 Borg Scale

   The Borg Scale represents a simple method to rate perceived exertion and can be compared to other scales, such as VAS. It is used for various purposes, such as measuring patient's exertion during a performance test or assessing the intensity of training and competition in athletes [30].

   The original scale developed by Borg ranging from 6 (no exertion at all) to 20 (maximal exertion) was updated and transformed into a combined category-ratio scale CR10 with the ratings 0 (nothing at all) to 10 (very very hard) [31, 32].

   The latter will be used in the present study. Subjects will be instructed to rate their work related physical exertion twice per day, at the end of the morning and in the late afternoon. The indicated Borg value should reflect how heavy and strenuous work feels to them considering all sensations of physical stress, effort and fatigue.

   2.4 Measurements

   2.4.1 Anthropometric measurements

   Anthropometric measurements include body height, body weight and waist circumference. Body height will be assessed without shoes by a medical measuring stick to the nearest mm. The measurement of body weight will be performed on subjects in light clothing without shoes by a medical scale with an accuracy of 0.1 kg.

   Waist circumference will be determined midway between the lowest rib and the iliac crest according to the Swiss Heart Foundation using a medical measuring tape with a precision of 0.1 cm. The measurement will be carried out on standing subjects after a moderate expiration.

   2.4.2 20-meter shuttle run

   The multistage 20-meter shuttle run is a common endurance fitness test to evaluate the maximal aerobic power of healthy adults [33]. It is simple in use and economical and large groups can be tested at once.

   This test will be conducted on a flat, non-slip surface and participants will be instructed to run back and forth between two lines, which are 20 meters apart (Figure 1). Running velocity is determined by intervals between two audio signals emitted by a pre-recorded tape. Subjects have to touch the 20 meter lines simultaneously with the sound of these signals. The initial running velocity is 8.5 km/h. Every minute (stage), the intervals are shortened and speed is increased by 0.5 km/h. The test ends when the subject gives up or when he can no longer keep the pace and does not reach the line in time (> 3 metre away from the 20 meter line) twice in a row.

   The test result corresponds to the number of reached stages. According to a validated table [34], this score is used to predict maximal oxygen uptake (VO2max), which can be compared to age-dependent normative data for males and females.

   Validity of the 1 minute stage version of the 20-meter shuttle run to predict VO2max in adults was established by Léger et al. [35], who compared the maximal shuttle run speed to VO2max attained during a multistage treadmill test.

   In addition, blood pressure and oxygen saturation will be assessed prior to testing in order to detect potential contraindications. Resting pulse and recovery pulse (2 minutes after test) will be measured and heart rate will be continuously recorded during test. Furthermore, participants will be instructed to rate their perceived physical exertion before and after test using the Borg scale.

   2.4.3 SenseWear Mini armband

   The SenseWear Mini armband is a small, lightweight and wireless multisensory activity monitor developed by Bodymedia (Pittsburgh, Pennsylvania, USA), which integrates motion data from a three-axis accelerometer along with several other physiological sensors such as heat flux, skin temperature and galvanic skin response. Validity was established by Johannsen et al. [36] comparing energy expenditure estimates of the SenseWear Mini armband against the criterion method 'Doubly-Labeled-Water' in healthy adults.

   The subjects will be instructed to wear the SenseWear Mini armband on the upper left arm (triceps area) for 7 consecutive days, including while sleeping, with the exception of one hour daily spent on personal hygiene (23 hours per day). Reliability of this assessment period has been previously shown [37].

   For recording non-wearing periods, such as water activities and showers, participants will be asked to keep a diary. The physiological data collected by the armband's sensors will be processed by specific algorithms (professional software V.7.0, algorithm V.2.2.4) to calculate participants' daily energy expenditure, METs, physical activity duration at different intensities and the number of steps. Gender, age, height, weight, smoking status and handedness will also be considered in these calculations.

   2.5 Statistical analysis

   Statistical analyses will be done using the software R (version 2.15.1) and IBM SPSS Statistics (version 19.0). Statistical significance will be acquired if a p value of less than 0.05 is attained.

   Data will be presented by descriptive statistics within occupational groups. Cross tables are reported as counts and percentages. Ordinal variables are reported as median and Interquartile range (IQR). Metric variables are reported as mean and standard deviation (SD).

   To evaluate primary endpoints, linear regressions will be performed. Independent variable is "occupational group", dependent variables are "average daily active energy expenditure", "average daily physical activity duration" and "average daily number of steps". Optionally, personal and job related factors can be included in the regression analyses as covariates. If appropriate, data will be log-transformed. Regression results will be presented as differences of means between "occupational categories" with corresponding 95% confidence intervals (C.I.) and p-values. In case of logarithmic distributed data, geometric mean ratios will be presented.

   To evaluate secondary endpoints, linear regressions will be conducted. In case of ordinal variables, non-parametric methods will be applied.

   Furthermore, the mean and individual time courses of physical activity periods will be plotted for all primary and secondary variables.

   2.6 Sample-size calculation

   Since "average daily active energy expenditure" measured by the SenseWear Mini armband represents a valid and reliable parameter, it is considered to be the most important primary endpoint of the present investigation. For this reason, only this variable is subject to a power calculation. In a previous study, the SD of "average daily active energy expenditure" during a normal work shift was found to be 730 kcal [38]. The expected mean difference between the three occupational groups will be around 500 kcal. Assuming a sample size of 100 subjects in each occupational group, there is a power of >90% to detect a mean difference of 500 kcal between any of these groups. This calculation is based on the assumption of a within group SD of 730 kcal and on a two-sided significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Full-time employment
* 18 to 65 years
* Sufficient knowledge of the German language

Exclusion Criteria:

* No consent for participation
* Movement restrictions
* Various diseases and accidents within the last three months
* Night shifts

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult full-time employees
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Average daily active energy expenditure during working time | 7 days
Average daily physical activity duration at different intensities during working time | 7 days
Average daily number of steps during working time | 7 days

SECONDARY OUTCOMES:
IPAQ: Total and subtotal domain specific scores (work, leisure-time, transport, domestic & garden [MET-min/week] and sitting time | 7 days
SF-36: Total and subtotal domain specific scores | 1 month
VAS: Scores of perceived work and leisure-time physical exertion and effort | 7 days
Results of the 20 meter shuttle run: predicted VO2max | 1 day
Results of the SenseWear Mini armband in recreation: activity and energy scores | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Jörg D Leuppi, Prof. MD PhD, Principal Investigator — Cantonal Hospital Baselland, Switzerland
Locations (1):
- Cantonal Hospital Baselland, Liestal, Liestal, Switzerland